CLINICAL TRIAL: NCT00769795
Title: Phase II Study of Neoadjuvant IMC-A12 Combined With Androgen Deprivation Prior to Prostatectomy
Brief Title: Study of Effectiveness of IMC-A12 Antibody Combined With Hormone Therapy Prior to Surgery to Treat Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Bruce Montgomery, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6857 (FH/UWCC ID); NIH P50 CA097186; 6857 (Other: FHCRC/UWMC Cancer Consortium)
Record Dates: First submitted 2008-10-07; First posted 2008-10-09 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostatic neoplasm; androgen deprivation therapy; insulin-like growth factor receptor I; neoadjuvant; prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cixutumumab; bicalutamide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): Bicalutamide 50 mg daily for 12 weeks Goserelin 10.8 mg SC once IMC-A12 10 mg/kg IV every three weeks for 12 weeks
  Interventions: Drug: IMC-A12; Drug: Bicalutamide; Drug: Goserelin

INTERVENTIONS:
Drug: IMC-A12 — IMC-A12 will be administered every 2 weeks for a total of 6 doses at 10 mg/kg per dose. The last dose of IMC-A12 will be at least 2 weeks prior to prostatectomy.
  Other Names: Cixutumumab
Drug: Bicalutamide — Bicalutamide 50 mg daily orally for 12 weeks
Drug: Goserelin — 10.8 mg subcutaneous once

SUMMARY:
The purpose of this study is to determine whether combination treatment of prostate cancer with IMC-A12 (an antibody which blocks insulin-like growth factor receptor activity) with hormonal therapy (testosterone lowering) before prostatectomy, will be more effective than prior results with hormonal therapy alone.

DETAILED DESCRIPTION:
Androgen deprivation has long been the principal means of controlling advanced prostate cancer, but it does not cure the disease and all patients ultimately progress if tumor is not eliminated with definitive local therapy. Neoadjuvant androgen deprivation prior to radical prostatectomy can downstage localized disease and reduce the likelihood of residual disease at the margins, but does not improve failure free survival. It has been demonstrated that despite androgen deprivation with luteinizing hormone releasing hormone (LHRH) agonists or orchiectomy, prostate tissue and prostate cancer maintain levels of androgens which are more than adequate to continue to stimulate the androgen receptor and downstream signaling. These levels of androgen may continue to allow both survival of tumor cells and induction of resistance by overexpression of receptor.

The anti-insulin-like growth factor type I receptor (IGF-IR) antibody IMC-A12 blocks translocation of the androgen receptor to the nucleus, dramatically augmenting efficacy of androgen deprivation in human prostate xenograft models. The combination of androgen deprivation with IMC-A12 is anticipated to more effectively treat cancer within the prostate, optimizing local control, while potentially eliminating micrometastatic disease. We propose to test this hypothesis in this phase II study, administering neoadjuvant androgen deprivation therapy IMC-A12 prior to radical prostatectomy for patients with clinically localized, high risk prostate cancer for 3 months.

Patients with clinically localized, and surgically resectable (cT1-T3) prostate cancer, at high risk for relapse who are candidates for radical prostatectomy will be treated with LHRH agonist and androgen receptor antagonist combined with IMC-A12, 10 mg/kg given intravenously every 14 days for 12 weeks. Patients will undergo biopsy of the prostate prior to treatment and radical prostatectomy 12 weeks after initiation of treatment.

The primary endpoint of the study is to evaluate the ability of LHRH agonist with IMC-A12 to induce a complete pathologic remission

Samples from the current study will be compared to control, untreated prostatectomy specimens from the Northwest Prostate SPORE Tissue Core and a concurrent set of specimens from patients treated with 12 weeks of combined androgen deprivation.

ELIGIBILITY:
Inclusion Criteria:

* Men 18 years or older with clinically localized prostate cancer who have chosen surgery (prostatectomy) and are at high risk of cancer relapse due to clinical stage, Gleason Score, PSA level, or a combination of the three.
* Good health and laboratory values within reasonable limits

Exclusion Criteria:

* Patients with prostate cancer that has spread outside the prostate.
* Patients who have low testosterone
* Patients who have received hormonal therapies or drugs which affect hormone metabolism
* Patients with serious medical conditions such as diabetes, other cancers, stroke, cardiovascular disease.
* Patients who are receiving other investigational therapy or chemotherapy.
* Patients who are unwilling to use contraceptives during and for a short time after the study
* Inability to give informed consent for any reason

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-10; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is to determine the effects of combining androgen deprivation with IMC-A12 on pathologic tumor stage (pathologic complete response). | At the time of prostatectomy after 3 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Montgomery, M.D., Principal Investigator — University of Washington and Seattle Cancer Care Alliance; James P Dean, M.D., Ph.D., Principal Investigator — University of Washington and Seattle Cancer Care Alliance; Stephen Plymate, M.D., Principal Investigator — University of Washington; John M Corman, MD, Principal Investigator — Virginia Mason Medical Center
Locations (3):
- United States (3):
  - Virginia Mason Medical Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Dean JP, Sprenger CC, Wan J, Haugk K, Ellis WJ, Lin DW, Corman JM, Dalkin BL, Mostaghel E, Nelson PS, Cohen P, Montgomery B, Plymate SR. Response of the insulin-like growth factor (IGF) system to IGF-IR inhibition and androgen deprivation in a neoadjuvant prostate cancer trial: effects of obesity and androgen deprivation. J Clin Endocrinol Metab. 2013 May;98(5):E820-8. doi: 10.1210/jc.2012-3856. Epub 2013 Mar 26. PMID 23533230